CLINICAL TRIAL: NCT01073189
Title: Effect of Combination Intra-Renal Infusion of Fenoldopam Mesylate and High Dose Diuretics on Peak Serum Creatinine and Incidence of Renal Replacement Therapy in Patients With Early Acute Kidney Injury
Brief Title: Intra-Renal Therapy of Diuretic Unresponsive Acute Kidney Injury
Acronym: IR-FTA
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: withdrew due to funding
Sponsor: Southeast Renal Research Institute (Other)
Responsible Party: James A. Tumlin MD Director Southeast Renal Research Institute, Southeast Renal Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IR-FTA
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Kidney Failures, Acute
Keywords: Acute kidney injury; Fenoldopam mesylate; Benephit catheter
MeSH Terms: conditions — Acute Kidney Injury | interventions — Fenoldopam; Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intra-Renal Fenoldopam (Experimental): Intra-Renal Fenoldopam: Patients randomized to this wing will undergo placement of Angiodynamics Benefit catheter and receive intra-renal infusion of fenoldopm mesylate
  Interventions: Drug: Intra-Renal Fenoldopam
- Diuretic Control (Active Comparator): Patients in the control group will be randomized to receive intra-venous diuretics as a comparator control
  Interventions: Drug: Furosemide

INTERVENTIONS:
Drug: Intra-Renal Fenoldopam — Placement of an intra-renal catheter for infusion of fenoldopam mesylate
  Other Names: Angiodynamics Benefit Catheter; Fenoldopam mesylate
  Arms: Intra-Renal Fenoldopam
Drug: Furosemide — Patients randomized to the Diuretic Control group will receive intravenous furosemide as an active control
  Other Names: Lasix
  Arms: Diuretic Control

SUMMARY:
Randomized prospective trial of patients with diuretic unresponsive acute kidney injury where patients will receive standard supportive therapy with diuretics versus intra-renal delivery of the vasodilator fenoldopam mesylate.

Patients with rising creatinine who fail to respond to bolus diuretics will be treated with a prolonged course of diuretics or undergo placement of a catheter within the renal arteries that allows for infusion of fenoldopam mesylate. The rational is that early delivery of a high dose vasodilator may reverse the decline of renal function in patients with severe acute kidney injury.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common complication of hospitalized patients and is associated with increased morbidity and mortality 1. The pathogenesis of AKI is a complex, time dependent process involving multiple variables including significant reductions in renal blood flow (RBF), interstitial infiltration by activated neutrophils and obstruction of tubule lumens with necrotic debris. In both human studies and animal models, the change in RBF is an early event with reductions in RBF between 40-50%. The mechanisms by which blood flow falls after the onset of AKI is unknown, but release of multiple vasoconstrictors coupled with a loss of autoregulation leads to prolonged reductions in RBF 2. The loss of the ability to vasodilate and autoregulate renal blood flow increases the sensitivity to additional ischemic and nephrotoxic insults.

Because reductions in RBF contribute to progression of AKI, clinical maneuvers that restore blood flow to ischemic kidneys offer the potential to significantly reduce patient mortality3. Consequently, numerous vasodilators have been investigated to determine whether restoring blood flow clinically to reduces the incidence of dialysis dependent AKI. Some agents including fenoldopam mesylate have shown encouraging results in specific sub-populations, but the benefits of other agents including atrial natriuretic peptide were offset by the development of systemic hypotension. The hypotenisve effects of these agents are a significant limitation to efforts to restore blood flow to ischemic kidneys. Moreover, the potential for additive hypotension and other side effects impedes the creation of "cocktails" of multiple agents which could have the ability to simultaneously activate numerous different protective pathways. Recent work using the FlowMedica Benephit catheter has shown that intra-renal delivery of vasodilators allows for targeted organ protection without the development of systemic side-effects. Moreover, the intra-renal delivery of fenoldopam mesylate and other vasodilators allows for supra-pharmacologic doses leading to and prolonged beneficial effects on RBF and GFR. We hypothesize that intra-renal delivery of fenoldopam mesylate to patients with early AKI will significantly reduce the number patients requiring renal replacement therapy. To investigate this hypothesis, we propose to study patients with "diuretic-resistant" AKI and randomize patients to supportive care with intermittent diuretics versus a 24 hour intra-renal infusion of fenoldopam mesylate in combination with intermittent diuretic therapy. The trial will be a randomized prospective, open-labeled study of 35 patients with early AKI defined as a 1.0 mg/dl rise in serum creatinine above baseline and/or two consecutive hours of urine output less than 20 mls/hr. The primary endpoint of the study will be peak serum creatinine at day #4 and the number of patients requiring renal replacement therapy or dying within 8 days of the onset of AKI. Additional data will be collected on the safety of implementation and the complications associated with a 24 hour infusion of fenoldopam using the Angiodynamics Benephit catheter

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  1. Any patient age 18 or over with a 1.0 mg/dl rise in serum Cr within 48 hours or a fall in urine output of less than 20 mls/min X 2 consecutive hours.

     AND one of the two following Options
  2. Failure to double urine output within two hours of a 1.5 mg/kg bolus Furosemide -OR-
  3. Failure to maintain a 50% increase in urine output for 4 consecutive hours following a single 1.5 mg/kg bolus of furosemide WITH an MD performed Urinalysis documenting the presence of 3 or more "muddy brown casts" per low powered field (LPF) or the presence of a "free renal tubular cells"

Exclusion Criteria:

* Exclusion Criteria:

  1. Patients with APACHE scores greater than 25 (or felt by the principle investigators not to survive more than 24 hours)
  2. Patients with a MAP < 65 on two or more vasopressor or any patient requiring 3 or more presser agents (nor epinephrine, + epinephrine or vasopressin) to maintain a MAP of 65 mm Hg .
  3. Patients receiving acute or chronic peritoneal or hemodialysis during current hospitalization
  4. Patients receiving dopamine or fenoldopam infusion within the previous 24 hours
  5. Patients requiring hemodynamic support with an intra-aortic balloon pump
  6. Patients with known HIV seropositivity
  7. Pregnant or lactating women
  8. Patients actively receiving NSAIDS or COX-2 antagonists
  9. Patients with history of uncontrolled cardiac arrhythmia
  10. Patients who cannot give informed consent.
  11. Patients with a known hypersensitivity to fenoldopam mesylate
  12. Patients with known bleeding diathesis
  13. Patients known blockage to one or more renal arteries
  14. Patients with known condition that would increase the likelihood of vascular perforation, trauma, or dissection such as Marfan's syndrome, cystic medial necrosis, abdominal or thoracoabdominal aortic dissection, mycotic aneurysm, abdominal aneurysm, thoracoabdominal aneurysm, renal artery aneurysm, thoracic aneurysm involving the visceral region of the aorta, and severe calcification in the area of the renal arteries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Peak creatinine at day 4 Renal replacement therapy at 8 days All-cause mortality at 21 days | Day 4, Day 8 and Day 21

SECONDARY OUTCOMES:
24 hour urinary volume at 72 hours Time to > 2.0 liters/24 hours Time to serum Cr < 2.5 mg/dl All cause mortality at 90 and 180 days | All cause mortality at 90 and 180 days

CONTACTS AND LOCATIONS:
Overall Officials: James A Tumlin, MD, Principal Investigator — Southeast Renal Research Institute
Locations (1):
- Erlanger Medical Center, Chattanooga, Tennessee, United States

REFERENCES:
- [Derived] Esezobor CI, Bhatt GC, Effa EE, Hodson EM. Fenoldopam for preventing and treating acute kidney injury. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD012905. doi: 10.1002/14651858.CD012905.pub2. PMID 39607014